CLINICAL TRIAL: NCT01260506
Title: Single-Arm Open-Label Multicenter Study of VB-111 in Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VB-111-122
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Glioblastoma Multiforme
Keywords: Relapsed Glioblastoma Multiforme, GBM
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VB-111 (Experimental): Antiangiogenic and vascular disruptive agent
  Interventions: Drug: VB-111; Drug: Bevacizumab

INTERVENTIONS:
Drug: VB-111
Drug: Bevacizumab — Upon progression, subjects will receive a combination therapy of VB-111 and standard of care bevacizumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of VB-111 in patients with Relapsed Glioblastoma Multiforme.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed diagnosis of glioblastoma multiforme or gliosarcoma;
2. Measurable disease by RANO criteria;
3. Disease progression or recurrence following standard of care treatment with temozolomide and radiation;
4. An interval of at least 4 weeks between prior surgical resection and study enrollment;
5. An interval of at least 12 weeks between prior radiotherapy or at least 4 weeks from prior chemotherapy, and enrollment in this protocol;
6. Recovered to Grade 1 or less from the toxic effects of any earlier intervention;
7. Karnofsky performance status > 60%

Exclusion Criteria:

1. Prior anti-angiogenic therapy including VEGF sequestering agents (ie bevacizumab, aflibercept, etc) or VEGFR inhibitors (cediranib, pazopanib, sunitinib, sorafenib, etc);
2. Prior stereotactic radiotherapy;
3. Active infection;
4. Evidence of CNS haemorrhage CTCAE grade 2 or above on baseline MRI;
5. Subjects who suffered from an acute cardiac event within the last 12 months;
6. Subjects with active vascular disease, either myocardial or peripheral;
7. Subjects with proliferative and/or vascular retinopathy;
8. Subjects with known active second malignancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2010-12; Primary Completion 2015-07-23 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From date of study entry until the date of death from any cause (up to 10 years)

SECONDARY OUTCOMES:
Progression Free Survival | 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Uthsc- Ctrc, San Antonio, Texas
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel